CLINICAL TRIAL: NCT05996185
Title: Phase II Study of Mogamulizumab With DA-EPOCH or CHOEP in Patients With Aggressive T-cell Lymphoma
Brief Title: Study of Mogamulizumab With DA-EPOCH or CHOEP in Patients With Aggressive T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Principal Investigator, Tarsheen Sethi, MD, MSCI, Assistant Professor of Medicine, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000037447; 000 (Other: CTGTY)
Record Dates: First submitted 2023-07-24; First posted 2023-08-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-04

CONDITIONS: T Cell Lymphoma; T-cell Lymphoma
Keywords: Relapsed; Refractory; Adult T-Cell Leukemia/Lymphoma; Cutaneous T-cell lymphoma; Mycosis Fungoides/Sézary syndrome; DA-EPOCH; Mogamulizumab; CHOEP
MeSH Terms: conditions — Lymphoma, T-Cell; Recurrence; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — mogamulizumab; EPOCH protocol; Doxorubicin; Cyclophosphamide; Vincristine; Prednisone; CHOEP protocol; Etoposide

STUDY DESIGN:
Intervention Model Description: All subjects are scheduled to receive six cycles of DA-EPOCH + Mogamulizumab
  Cycle 1: Mogamulizumab on days 1,8,15, of a 21-day cycle with DA-EPOCH on day 1.
  Cycles 2 to 6: Mogamulizumab on day 1 with DA-EPOCH or CHOEP
Masking Description: Selection of regimen will be at the treating investigator's discretion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mogamulizumab + DA-EPOCH or CHOEP (Experimental): All subjects are scheduled to receive six cycles of DA-EPOCH + Mogamulizumab
  Cycle 1: Mogamulizumab on days 1,8,15, of a 21-day cycle with DA-EPOCH on day 1.
  Cycles 2 to 6: Mogamulizumab on day 1 with DA-EPOCH or CHOEP
  Mogamulizumab will be administered modified to a 21-day cycle in combination with chemotherapy. Subjects will receive 1.0 mg/kg of mogamulizumab as an IV infusion over at least 1 hour on Days 1, 8, 15 of the first cycle and Day 1 for the subsequent cycles. This is based on prior studies with mogamulizumab in combination of chemotherapy.(15) This dosing regimen will ensure the first 4 doses are given weekly at a dose of 1 mg/kg. Subsequent dosing on a 21-day schedule to coincide with the frequency of administration of DA-EPOCH or CHOEP to allow for simpler co-administration of the study drugs. In addition, this study proposes to leverage the immunomodulatory role of mogamulizumab, the dosing for this has not been previously established or explored.
  Interventions: Drug: Mogamulizumab; Drug: DA-EPOCH Protocol; Drug: CHOEP protocol

INTERVENTIONS:
Drug: Mogamulizumab — Mogamulizumab is a defucosylated, humanized, monoclonal antibody (Mab) with enhanced antibody dependent cellular cytotoxicity that binds to CCR4. The lack of fucose results in the antibody eliciting more potent ADCC than conventionally produced antibodies. Mogamulizumab is devoid of complement dependent cytotoxicity.
  CC Chemokine receptor 4 is over expressed on the surfaces of cells comprising several T-cell malignancies such as peripheral T-cell lymphoma (PTCL) and CTCL and is a potential target for anti-neoplastic therapy in these disorders.
  Other Names: Poteligeo
Drug: DA-EPOCH Protocol — EPOCH is an intensive chemotherapy regimen intended for treatment of aggressive non-Hodgkin's lymphoma.
  Other Names: dose-adjusted etoposide, doxorubicin, and cyclophosphamide with vincristine and prednisone
Drug: CHOEP protocol — CHOEP is an intensive chemotherapy intended for treatment of aggressive t-cell lymphoma.
  Other Names: dose-adjusted Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Etoposide, Prednisone

SUMMARY:
Single-arm Phase II study evaluating the combination of mogamulizumab (MOGA) added on top of standard of care dose adjusted EPOCH (DA-EPOCH) or CHOEP in patients with newly diagnosed or relapsed/refractory (for CTCL only) aggressive T-cell lymphoma including patients with Adult T-cell leukemia/lymphoma (ATLL).

DETAILED DESCRIPTION:
This is a single arm, open label, multicenter phase II study of DA-EPOCH or CHOEP and Mogamulizumab in patients with newly diagnosed or relapsed/refractory (for CTCL only) aggressive T-cell lymphomas including ATLL and transformed Mycosis Fungoides/Sézary syndrome (MF/SS). The investigators hypothesize that this combination is effective and will produce a CR rate that is statistically larger than 40%, a rate based on historical data from the current standard of care. DA-EPOCH or CHOEP and Mogamulizumab will be administered for 6 cycles and depending on the histology, consolidative strategies including SCT will be considered. Response assessments will occur at pre-specified intervals. Dose adjustments for specific toxicities with drugs are detailed in the protocol. Based on statistical analysis, a maximum of 22 patients will need to be accrued to obtain a sample of 19 evaluable patients for disease response.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of T-cell Non-Hodgkin lymphoma (TNHL) will be enrolled in this study.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 unless compromised by lymphoma with anticipated benefit from chemotherapy as determined and documented by the investigator.
3. Histologically confirmed T-cell Non-Hodgkin lymphoma (T-NHL), including but not limited to:

   * Peripheral T-cell lymphoma not otherwise specified (PTCL nos)
   * Angioimmunoblastic T-cell lymphoma (AITL)
   * Anaplastic large-cell lymphoma (ALCL)
   * Cutaneous T-cell lymphoma (CTCL), including mycosis fungoides (MF)/sezary syndrome patients for whom multi-agent chemotherapy is indicated
   * Transformed mycosis fungoides/Sézary syndrome
   * Enteropathy-associated T-cell lymphoma (EATL)
   * Subcutaneous panniculitis-like T-cell lymphoma (SCPTCL)
   * Hepatosplenic T- cell lymphomas
   * Gamma delta T-cell lymphomas
   * Adult T-cell lymphoma leukemia (ATLL)
   * T-prolymphocytic leukemia with nodal or visceral involvement
4. Prior therapy- patients with aggressive T-cell lymphoma may have received one cycle of CHOP, CHOEP or EPOCH before enrollment, if necessary, to control the disease.
5. For patients with peripheral T-cell lymphoma (PTCL): At least one measurable target lesion ≥ 1.5 cm
6. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   * Not a woman of childbearing potential (WOCBP) as defined in Appendix 4 OR
   * A woman of childbearing potential (WOCBP) - see Appendix 4 for definition of WOCBP - must have a negative serum or urine pregnancy test during screening and must agree to follow instructions for using acceptable contraception (Appendix 5) from the time of signing consent, and at least 180 days (6 months) after her final dose of mogamulizumab.
7. A male patient must agree to use a contraception as detailed in Appendix 5 of this protocol during the treatment period and for at least at least 180 days (6 months) after her final dose of mogamulizumab and refrain from donating sperm during this period.
8. Adequate organ and bone marrow function resulted ≤ 10 days prior to first dose of protocol-indicated treatment unless compromised by disease involvement of bone marrow, spleen, or liver as determined and documented by the investigator.
9. Patients previously treated with anti-CD4 antibody or alemtuzumab are eligible provided their CD4+ cell counts are ≥ 200/mm.

Exclusion Criteria:

1. Has received prior systemic anti-cancer therapy including investigational agents ≤ 3 weeks prior to first dose of study treatment on Cycle 1, Day 1. Skin directed treatments, including topicals and radiation within 2 weeks of study treatment. However, patients with rapidly progressive malignant disease may be enrolled prior to this period after discussion with the sponsor investigator.
2. Has received radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
3. If patient received major surgery, participants must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Patients on any immunomodulatory drug for concomitant or intercurrent conditions other than T-cell lymphoma or who have received any of these agents within 4 weeks of treatment, including but not limited to the following, will be excluded: low dose or oral methotrexate; azathioprine; iv immunoglobulin; low dose or oral cyclophosphamide; cyclosporine; mycophenolate; infliximab; etanercept; leflunomide; adalimumab; lenalidomide; abatacept; rituximab; anakinra; interferon-β IL-2 and natalizumab. . Concurrent use of topical steroids or therapies for CTCL is allowed as indicated in the protocol.
5. Pregnant or breast-feeding females. A WOCBP who has a positive urine pregnancy test within 72 hours of treatment start. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
6. Has received a live vaccine within 30 days prior to the first dose of study drug.

   Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg,FluMist®) are live attenuated vaccines and are not allowed.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
8. Active uncontrolled infection requiring systemic therapy (patients must be afebrile for ≥ 48 hours and off antibiotics prior to treatment). If fever is attributed to tumor fever (B symptom) then these criteria would not apply.
9. Active myocarditis, regardless of etiology; or New York Heart Association (NYHA) functional classification III-IV heart failure (Appendix 4).
10. Known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided participants are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
11. Diagnosed with a malignancy, not treated under the study (hormonal therapy for breast or prostate cancer excepted), in the past 2 years. However, patients with nonmelanoma skin cancers, melanoma in situ, localized cancer of the prostate with current prostate-specific antigen of < 0.1 ng/mL, treated thyroid cancer or cervical carcinoma in situ or ductal/lobular carcinoma in situ of the breast with in the past 2 years may enroll as long as there is no current evidence of disease.
12. Known severe hypersensitivity (≥Grade 3) to mogamulizumab and/or any of its excipients and /or EPOCH/or CHOEP or any of its excipients.
13. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
15. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Prior allogeneic stem cell transplant within last 2 years or active graft vs. host disease (GVHD).
18. Known active autoimmune disease will be excluded if the disease requires active medical treatment. (For example, Graves' disease; systemic lupus erythematosus; rheumatoid arthritis; Crohn's disease; psoriasis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Complete response after 6 cycles of treatment with the combination Mogamulizumab and standard of care DA-EPOCH or CHOEP | 6 cycles (126 Days)
  As assessed by the Lugano criteria for PTCL(16) and the global response score for CTCL(17)

SECONDARY OUTCOMES:
Occurrence of toxicity | 2 years
  using the NCI Common Terminology Criteria for Adverse Events version 5 (CTCAE v5) for grading.
Progression free survival (PFS) | 2 years
  Defined as the time from enrollment to earliest of progression, death or follow-up
Overall survival (OS) | 2 years
  defined as time from the time from enrollment to earlier of death or last follow-up
Duration of response | 2 Years
  (including both scenarios -censored at the time of subsequent therapy without disease progression, such as stem cell transplant and total duration including after SCT)
Time to best response | 2 years
  Defined as the time from treatment initiation to best response
Overall response rate | 2 years
  Defined as the percentage of patients whose cancer shows a partial response or complete response

CONTACTS AND LOCATIONS:
Overall Officials: Tarsheen Sethi, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Cancer Center, Clinical Trials Office, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] Bazarbachi A, Suarez F, Fields P, Hermine O. How I treat adult T-cell leukemia/lymphoma. Blood. 2011 Aug 18;118(7):1736-45. doi: 10.1182/blood-2011-03-345702. Epub 2011 Jun 14. PMID 21673346
- [Background] Ellin F, Landstrom J, Jerkeman M, Relander T. Real-world data on prognostic factors and treatment in peripheral T-cell lymphomas: a study from the Swedish Lymphoma Registry. Blood. 2014 Sep 4;124(10):1570-7. doi: 10.1182/blood-2014-04-573089. Epub 2014 Jul 8. PMID 25006130
- [Background] Horwitz S, O'Connor OA, Pro B, Illidge T, Fanale M, Advani R, Bartlett NL, Christensen JH, Morschhauser F, Domingo-Domenech E, Rossi G, Kim WS, Feldman T, Lennard A, Belada D, Illes A, Tobinai K, Tsukasaki K, Yeh SP, Shustov A, Huttmann A, Savage KJ, Yuen S, Iyer S, Zinzani PL, Hua Z, Little M, Rao S, Woolery J, Manley T, Trumper L; ECHELON-2 Study Group. Brentuximab vedotin with chemotherapy for CD30-positive peripheral T-cell lymphoma (ECHELON-2): a global, double-blind, randomised, phase 3 trial. Lancet. 2019 Jan 19;393(10168):229-240. doi: 10.1016/S0140-6736(18)32984-2. Epub 2018 Dec 4. PMID 30522922
- [Background] Mehta N, Maragulia JC, Moskowitz A, Hamlin PA, Lunning MA, Moskowitz CH, Zelenetz A, Matasar MJ, Sauter C, Goldberg J, Horwitz SM. A retrospective analysis of peripheral T-cell lymphoma treated with the intention to transplant in the first remission. Clin Lymphoma Myeloma Leuk. 2013 Dec;13(6):664-70. doi: 10.1016/j.clml.2013.07.005. Epub 2013 Sep 11. PMID 24035712
- [Background] Maeda Y, Nishimori H, Yoshida I, Hiramatsu Y, Uno M, Masaki Y, Sunami K, Masunari T, Nawa Y, Yamane H, Gomyo H, Takahashi T, Yano T, Matsuo K, Ohshima K, Nakamura S, Yoshino T, Tanimoto M. Dose-adjusted EPOCH chemotherapy for untreated peripheral T-cell lymphomas: a multicenter phase II trial of West-JHOG PTCL0707. Haematologica. 2017 Dec;102(12):2097-2103. doi: 10.3324/haematol.2017.167742. Epub 2017 Sep 29. PMID 28971899
- [Background] Toriyama E, Imaizumi Y, Taniguchi H, Taguchi J, Nakashima J, Itonaga H, Sato S, Ando K, Sawayama Y, Hata T, Fukushima T, Miyazaki Y. EPOCH regimen as salvage therapy for adult T-cell leukemia-lymphoma. Int J Hematol. 2018 Aug;108(2):167-175. doi: 10.1007/s12185-018-2455-x. Epub 2018 Apr 12. PMID 29651666
- [Background] Kim YH, Bagot M, Pinter-Brown L, Rook AH, Porcu P, Horwitz SM, Whittaker S, Tokura Y, Vermeer M, Zinzani PL, Sokol L, Morris S, Kim EJ, Ortiz-Romero PL, Eradat H, Scarisbrick J, Tsianakas A, Elmets C, Dalle S, Fisher DC, Halwani A, Poligone B, Greer J, Fierro MT, Khot A, Moskowitz AJ, Musiek A, Shustov A, Pro B, Geskin LJ, Dwyer K, Moriya J, Leoni M, Humphrey JS, Hudgens S, Grebennik DO, Tobinai K, Duvic M; MAVORIC Investigators. Mogamulizumab versus vorinostat in previously treated cutaneous T-cell lymphoma (MAVORIC): an international, open-label, randomised, controlled phase 3 trial. Lancet Oncol. 2018 Sep;19(9):1192-1204. doi: 10.1016/S1470-2045(18)30379-6. Epub 2018 Aug 9. PMID 30100375
- [Background] Zinzani PL, Karlin L, Radford J, Caballero D, Fields P, Chamuleau ME, d'Amore F, Haioun C, Thieblemont C, Gonzalez-Barca E, Garcia CG, Johnson PW, van Imhoff GW, Ng T, Dwyer K, Morschhauser F. European phase II study of mogamulizumab, an anti-CCR4 monoclonal antibody, in relapsed/refractory peripheral T-cell lymphoma. Haematologica. 2016 Oct;101(10):e407-e410. doi: 10.3324/haematol.2016.146977. Epub 2016 Jul 14. No abstract available. PMID 27418646
- [Background] Jo T, Matsuzaka K, Shioya H, Tominaga H, Sakai T, Kaneko Y, Hayashi S, Matsuo M, Taguchi J, Abe K, Shigematsu K, Kubota-Koketsu R. Mogamulizumab Plus EPOCH Therapy for Patients With Newly Diagnosed Aggressive Adult T-cell Leukemia/lymphoma. Anticancer Res. 2020 Sep;40(9):5237-5243. doi: 10.21873/anticanres.14527. PMID 32878812
- [Background] Ishida T, Jo T, Takemoto S, Suzushima H, Uozumi K, Yamamoto K, Uike N, Saburi Y, Nosaka K, Utsunomiya A, Tobinai K, Fujiwara H, Ishitsuka K, Yoshida S, Taira N, Moriuchi Y, Imada K, Miyamoto T, Akinaga S, Tomonaga M, Ueda R. Dose-intensified chemotherapy alone or in combination with mogamulizumab in newly diagnosed aggressive adult T-cell leukaemia-lymphoma: a randomized phase II study. Br J Haematol. 2015 Jun;169(5):672-82. doi: 10.1111/bjh.13338. Epub 2015 Mar 2. PMID 25733162
- [Background] Wilson WH, Grossbard ML, Pittaluga S, Cole D, Pearson D, Drbohlav N, Steinberg SM, Little RF, Janik J, Gutierrez M, Raffeld M, Staudt L, Cheson BD, Longo DL, Harris N, Jaffe ES, Chabner BA, Wittes R, Balis F. Dose-adjusted EPOCH chemotherapy for untreated large B-cell lymphomas: a pharmacodynamic approach with high efficacy. Blood. 2002 Apr 15;99(8):2685-93. doi: 10.1182/blood.v99.8.2685. PMID 11929754
- [Background] Ishida T, Joh T, Uike N, Yamamoto K, Utsunomiya A, Yoshida S, Saburi Y, Miyamoto T, Takemoto S, Suzushima H, Tsukasaki K, Nosaka K, Fujiwara H, Ishitsuka K, Inagaki H, Ogura M, Akinaga S, Tomonaga M, Tobinai K, Ueda R. Defucosylated anti-CCR4 monoclonal antibody (KW-0761) for relapsed adult T-cell leukemia-lymphoma: a multicenter phase II study. J Clin Oncol. 2012 Mar 10;30(8):837-42. doi: 10.1200/JCO.2011.37.3472. Epub 2012 Feb 6. PMID 22312108
- [Background] Yamamoto K, Utsunomiya A, Tobinai K, Tsukasaki K, Uike N, Uozumi K, Yamaguchi K, Yamada Y, Hanada S, Tamura K, Nakamura S, Inagaki H, Ohshima K, Kiyoi H, Ishida T, Matsushima K, Akinaga S, Ogura M, Tomonaga M, Ueda R. Phase I study of KW-0761, a defucosylated humanized anti-CCR4 antibody, in relapsed patients with adult T-cell leukemia-lymphoma and peripheral T-cell lymphoma. J Clin Oncol. 2010 Mar 20;28(9):1591-8. doi: 10.1200/JCO.2009.25.3575. Epub 2010 Feb 22. PMID 20177026
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Connor AM, Moshiri F. Advancement genioplasty: an important part of combination surgery in black American patients. Am J Orthod Dentofacial Orthop. 1988 Feb;93(2):92-8. doi: 10.1016/0889-5406(88)90285-5. No abstract available. PMID 3422534
- [Background] Trnavska Z, Trnavsky K, Kuhn K. [Effect of sodium salicylate on the metabolism of collagen proteins]. Fysiatr Revmatol Vestn. 1968 Dec;46(6):341-7. No abstract available. Czech. PMID 5749831
- [Background] Keinert K. [Experience with the cytological puncture of lymphographically stained lymph nodes in various regions]. Radiol Diagn (Berl). 1972;13(5):680-1. No abstract available. German. PMID 4656023
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564